CLINICAL TRIAL: NCT07337798
Title: Effects of Implementing Evidence-Based Clinical Nutrition Practice Guidelines in Surgical Intensive Care Units: A Cohort Study
Brief Title: Implementation of Clinical Nutrition Practice Guidelines in Surgical ICUs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: iPARIHS-SICU-2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: ICU Patients; Surgical; Nutrition Intervention; Enteral Nutrition; Enteral Nutrition Intolerance
Keywords: Clinical Nutrition; Surgical Intensive Care Units; i-PARIHS Framework; Implementation Science; Clinical practice guideline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guideline Implementation Group (Experimental): Participants in this single-arm study will receive an evidence-based, context-adapted clinical nutrition practice guideline implemented in surgical intensive care units (ICUs) using an i-PARIHS-guided translation strategy. The implementation includes guideline localization, expert consensus validation, education and training, on-site facilitation, audit and feedback, and continuous process optimization. Outcomes will be assessed before and after guideline implementation to evaluate changes in healthcare professional adherence to clinical nutrition recommendations and nutrition-related clinical outcomes among surgical critically ill patients.
  Interventions: Behavioral: Guideline Implementation

INTERVENTIONS:
Behavioral: Guideline Implementation — This behavioral intervention consists of the implementation of an evidence-based, context-adapted clinical nutrition practice guideline in surgical intensive care units (ICUs), guided by the integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework. The intervention includes systematic guideline selection based on existing surgical and critical care nutrition guidelines, contextual adaptation to the Chinese healthcare setting, guideline localization and expert consensus validation, and structured implementation strategies.
  Key components of the intervention include education and training of ICU healthcare professionals, on-site facilitation, audit and feedback, and continuous process optimization to support adherence to guideline recommendations. The intervention is delivered at the unit level and integrated into routine clinical practice in surgical ICUs. Outcomes are evaluated using a pre- and post-implementation design to assess changes in healt

SUMMARY:
The goal of this interventional clinical trial is to evaluate whether the implementation of an evidence-based, context-adapted clinical nutrition practice guideline can improve clinical nutrition management in surgical intensive care units (ICUs) in China. The guideline is selected based on the best available evidence from existing surgical and critical care nutrition guidelines, adapted to the Chinese healthcare context, and implemented using an i-PARIHS-guided translation strategy. The trial involves ICU healthcare professionals working in surgical ICUs of tertiary general hospitals, while assessing nutrition-related clinical outcomes among surgical critically ill patients.

The main questions it aims to answer are:

Does guideline implementation improve ICU healthcare professionals' adherence to recommended clinical nutrition practice guidelines?

Does the implementation of the clinical nutrition practice guideline improve the proportion of surgical critically ill patients who achieve recommended energy and protein intake targets during ICU stay?

Researchers will compare outcomes before and after guideline implementation to determine whether the i-PARIHS-guided guideline translation improves nutrition management processes, healthcare professional performance, and patient-related clinical outcomes.

Participants will:

Complete baseline and post-implementation assessments related to clinical nutrition knowledge, attitudes, and practices.

Participate in guideline-based education, training, and implementation activities guided by the i-PARIHS framework.

Apply the adapted clinical nutrition practice guideline during routine clinical care in surgical ICUs.

Be evaluated through on-site audits, questionnaires, and clinical data collection during the implementation process.

DETAILED DESCRIPTION:
This study is an interventional, multicenter implementation clinical trial designed to translate and apply an evidence-based clinical nutrition practice guideline in surgical intensive care units (ICUs) in China, guided by the i-PARIHS framework. The guideline is developed through a structured process that includes identification of best available evidence from existing surgical and critical care nutrition guidelines, contextual adaptation to the Chinese healthcare setting, guideline item localization, and expert consensus validation.

The implementation strategy is informed by the i-PARIHS framework, with particular emphasis on facilitation, local context assessment, and engagement of key stakeholders. A series of structured implementation activities, including education, training, on-site facilitation, audit and feedback, and continuous process optimization, are conducted to support guideline uptake in routine clinical practice. The implementation process follows a pre- and post-implementation design, allowing for comparison of outcomes before and after guideline translation.

The primary outcomes focus on (1) adherence of ICU healthcare professionals to recommended clinical nutrition practice guidelines and (2) the proportion of surgical critically ill patients achieving recommended energy and protein intake targets during ICU stay.

Secondary outcomes are assessed to comprehensively evaluate the impact of guideline implementation on nutrition delivery processes and patient-related clinical outcomes. These include:

Timing of enteral nutrition initiation after ICU admission

Frequency of enteral nutrition interruptions during ICU stay

Global Leadership Initiative on Malnutrition (GLIM) classification at ICU discharge

Cumulative daily energy and protein balance, including total caloric and protein surplus or deficit per day during ICU stay

Laboratory indicators at ICU discharge, including urea-to-creatinine ratio, serum albumin, globulin, interleukin-6 (IL-6), and C-reactive protein (CRP)

Length of ICU stay

Clinical outcomes during ICU hospitalization

All-cause 28-day mortality

Data are collected through a combination of on-site clinical audits, standardized questionnaires, electronic medical record extraction, and laboratory testing. Outcomes related to healthcare professionals are measured using structured adherence assessment tools and knowledge-attitude-practice evaluations, while patient-related outcomes are derived from routinely collected clinical and laboratory data.

The feasibility, appropriateness, and effectiveness of the guideline implementation are evaluated based on changes in outcome measures, process indicators, and participant satisfaction. The findings of this study are intended to inform scalable and context-sensitive strategies for optimizing clinical nutrition management in surgical ICUs within the Chinese healthcare system.

ELIGIBILITY:
Inclusion Criteria:

For ICU healthcare professionals:

Employed at one of the participating study sites (tertiary general hospitals)

Holds a valid Registered Nurse license issued in the People's Republic of China

Currently working in frontline clinical nursing care in a surgical intensive care unit (ICU) during the study period

At least 1 year of clinical working experience

Able to understand the study objectives and procedures

Willing to participate and able to provide written informed consent

For surgical critically ill patients (outcome assessment population):

Aged 18 years or older

Admitted to a surgical ICU due to surgical-related conditions, including trauma, infection, malignancy, or postoperative complications

Expected length of stay in the surgical ICU of at least 48 hours

No restriction on sex

Patient or legally authorized representative able to provide written informed consent

Exclusion Criteria:

For ICU healthcare professionals:

Currently pregnant, breastfeeding, or planning pregnancy during the study period

Temporarily assigned, rotating, externally dispatched, on long-term training, or on leave during the study period, making continuous participation impossible

Participation in other interventional studies that may interfere with the implementation of this study

Determined by the research team to have cognitive, communication, or other conditions that would make participation inappropriate

For surgical critically ill patients:

Diagnosed with brain death or awaiting organ donation

Pregnant or breastfeeding women

Concurrent participation in other nutrition-related clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence of ICU Healthcare Professionals to Clinical Nutrition Practice Guidelines | At baseline (prior to implementation) and at 6 months after implementation.
  Adherence of ICU healthcare professionals to clinical nutrition practice guidelines, assessed using structured audit tools based on key guideline recommendations, including nutrition assessment, initiation and delivery of nutrition support, monitoring, and documentation practices.

SECONDARY OUTCOMES:
Proportion of Surgical Critically Ill Patients Achieving Energy and Protein Intake Targets During ICU Stay | From ICU admission (Day 1) to ICU discharge
  The proportion of surgical critically ill patients whose actual daily energy and protein intake meets guideline-recommended targets during ICU stay. Energy and protein intake will be calculated based on prescribed targets and recorded enteral and/or parenteral nutrition delivery. Patients achieving both energy and protein targets will be considered as meeting the outcome.

OTHER OUTCOMES:
Time to Initiation of Enteral Nutrition After ICU Admission | From ICU admission (Day 1) to initiation of enteral nutrition (up to 7 days).
  Time from ICU admission to the initiation of enteral nutrition, measured in hours, based on medical records and nutrition orders.
Frequency of Enteral Nutrition Interruptions During ICU Stay | From ICU admission (Day 1) to ICU discharge
  Number of enteral nutrition interruption events per patient during ICU stay, including interruptions due to procedures, intolerance, or clinical decisions, as documented in medical and nursing records.
GLIM Classification | At ICU admission (Day 1) and ICU discharge
  Nutritional status at ICU admission and ICU discharge assessed using the Global Leadership Initiative on Malnutrition (GLIM) criteria, categorized according to standard GLIM diagnostic classifications.
Cumulative energy balance during ICU stay | From ICU admission (Day 1) to ICU discharge
  Cumulative energy balance was calculated as the sum of the daily differences between delivered energy intake and prescribed energy targets during the ICU stay.
Cumulative protein balance during ICU stay | From ICU admission (Day 1) to ICU discharge
  Cumulative protein balance was calculated as the sum of the daily differences between delivered protein intake and prescribed protein targets during the ICU stay.
Urea-to-Creatinine Ratio | At ICU admission (Day 1) and ICU discharge
  Serum urea-to-creatinine ratio measured at ICU admission (Day 1) and ICU discharge, derived from routine laboratory testing.
Serum Albumin Levels | At ICU admission (Day 1) and ICU discharge
  Serum albumin concentrations measured at ICU admission (Day 1) and ICU discharge based on routine laboratory tests.
Serum C-Reactive Protein (CRP) Level | At ICU admission (Day 1) and ICU discharge
  The serum CRP level will be measured from blood samples collected at ICU admission (Day 1) and ICU discharge. CRP is an acute-phase protein that reflects systemic inflammation. The measurement will be performed using standard laboratory methods available at the hospital laboratory. Data will be reported in mg/L.
Length of ICU Stay | From ICU admission (Day 1) to ICU discharge
  Duration of ICU hospitalization, measured in days from ICU admission to ICU discharge.
Clinical Outcomes During ICU Stay | From ICU admission(Day 1) to ICU discharge
  Clinical outcomes during ICU stay, including occurrence of major complications and need for advanced organ support, extracted from electronic medical records.
All-Cause 28-Day Mortality | Up to 28 days after ICU admission
  All-cause mortality within 28 days after ICU admission, determined from hospital records and follow-up data.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The study involves sensitive clinical and professional information collected from ICU healthcare professionals and critically ill patients, and the data are derived from routine clinical records across multiple centers. Due to privacy protection, data confidentiality requirements, and institutional data governance policies, individual-level data cannot be made publicly available.